CLINICAL TRIAL: NCT02063204
Title: An Open Label Comparative Study of the Pharmacokinetics, Safety and Tolerability of Selumetinib (AZD6244, ARRY 142886) (Hyd Sulfate) Following a Single Oral Dose in Subjects With Renal Impairment and Healthy Subjects
Brief Title: To Assess the Pharmacokinetics, Safety and Tolerability of Selumetinib in Renal Impaired Subjects and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00081
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumours
Keywords: Phase I, healthy, pharmacokinetics, renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HV selumetinib Stage 1 (Experimental): Healthy volunteer (HV)group to receive selumetinib 50mg (2x25mg) orally
  Interventions: Drug: selumetinib
- ESRD selumetinib Stage 1 (Experimental): End stage renal disease (ESRD)patients to recieve selumetinib 50mg (2x25mg) orally
  Interventions: Drug: selumetinib
- Selumetinib stage 2 (Experimental): If deemed necessary patients with mild and/or moderate and/or severe renal impairment will recieve selumetinib 50mg(2x25mg) orally
  Interventions: Drug: selumetinib

INTERVENTIONS:
Drug: selumetinib — selumetinib 50 mg (2x25mg) administered by mouth as capsules

SUMMARY:
A study to assess the pharmacokinetics, safety and tolerability of Selumetinib (AZD6244, ARRY-142886) in subjects with renal impairment and healthy subjects

DETAILED DESCRIPTION:
An open label study to assess the pharmacokinetics, safety and tolerability of 50 mg single oral dose of Selumetinib (AZD6244, ARRY-142886) in subjects with renal impairment and healthy subjects

ELIGIBILITY:
Inclusion Criteria all participants:

1. Male and female (non childbearing potential) subjects aged 18 years or more with suitable veins for cannulation or repeated venipuncture.
2. Have a weight of at least 50 kg (110 lbs) and body mass index (BMI) between 18 and 40 kg/m2, inclusive.

   Inclusion healthy volunteers only:
3. Must be in good health as determined by a medical history, physical examination, 12 lead ECG, clinical laboratory evaluations, and an ophthalmic examination performed before the administration of the investigational product.

   Inclusion renal impaired patients only:
4. Stable renal function

Exclusion Criteria all participants:

1. Subjects of Japanese or non Japanese Asian ethnicity.
2. Any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian (e.g. China, Taiwan, Korea, Philippines, Thailand, Vietnam and Malaysia). Asian Indians are acceptable.
3. Subjects who smoke more than 10 cigarettes or the equivalent in tobacco per day
4. In the opinion of the investigator, any evidence of additional severe or uncontrolled systemic disease (eg, currently unstable or uncompensated hepatic, cardiovascular, or respiratory disease) or laboratory finding, physical examination, hematology, clinical chemistry, urinalysis, vital signs, or 12-lead ECG that makes it undesirable for the subject to participate in the study.

   Exclusion renal impaired patients only:
5. Subjects with an active renal transplant (subjects who have previously received a renal transplant and are currently undergoing dialysis due to transplant failure may be enrolled).
6. Acute coronary syndrome within 6 months prior to administration of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic(PK) profile in terms of maximum observed plasma concentration (Cmax) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of area under plasma concentration-time curve from zero extrapolated to infinity (AUC) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of area under plasma concentration-time curve to time of last measurable concentration (AUC[0-t]) for selumetinib if AUC is not reportable in more than 80% of subjects | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, physical examinations, ophthalmologic assessments, vital signs, clinical laboratory assessments and 12-lead electrocardiograms. | From screening until follow up. Approximately 6 weeks for healthy volunteers and 8 weeks for renal patients
Description of the PK profile in terms of time to reach maximum observed concentration administration (tmax) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of area under the plasma concentration time curve from zero to 12 hours postdose (AUC[0-12]) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h, and12h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of terminal rate constant (λz), terminal elimination half-life (t1/2), apparent oral clearance (CL/F) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of apparent volume of distribution at steady state (Vss/F) and apparent volume of distribution during the terminal phase (Vz/F) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of mean residence time (MRT) and fraction unbound (fu), free Cmax (Cmax, u), free AUC (AUCu), free AUC(0-t) (AUC[0-t],u) and unbound CL/F (CL/Fu) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  This will be taken at visit 2 for Healthy volunteers and at visit 2 and 3 for patients with end stage renal disease
Description of PK profile in terms of the amount of drug excreted in urine (Ae) the fraction of dose excreted in urine (fe), renal clearance (CLR) for selumetinib and AUC, Cmax, tmax, t1/2, λz, AUC(0-12) and AUC(0-t) | The urine collection intervals will be from -12 to 0 (predose), and 0 to 6, 6 to 12, 12 to 24, 24 to 36, 36 to
  These collection will be taken on visit 2 for the healthy volunteers and on visit 2 and 3 if the patients can produce urine
Description of the PK profile in terms of the metabolite to parent AUC and Cmax ratios (MRAUC and MRCmax) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
  These samples will be taken on visit 2 for the healthy volunteers and on both visit 2 and visit 3
Description of the PK profile in terms of Ae, fe, and CLR for N-desmethyl selumetinib (and the amide metabolite, if deemed appropriate) | Samples taken at predose, 30min, 1h, 1h30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h,6h,7h,8h,12h,18h,24h,36h,48h and 76h
Description of the PK profile in terms of time-matched area under the plasma concentration time curve from 1 to 5 hours postdose (AUC[1-5]) | Sample taken predose, at 1h just before dialyse and at 5h after the end of the dialyse
  This will only be taken at the visit when dose is given 1h before dialyse start
Description of the PK profile in terms of cumulative amount extracted during dialysis (Ad[1-5]), and dialysis clearance (CLD) | Samples taken from dialysate collections over 1 hour intervals throughout the entire (approximately 4 hours) dialysis period ie, 0 to 1, 1 to 2, 2 to 3, 3
  This will only be collected during visit 2 and only on end stage renal disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Centre, US; Ian Smith, MD, Study Director — Astrazeneca United kingdom
Locations (1):
- Research Site, Orlando, Florida, United States

REFERENCES:
- See also: CSR_Synopsis_D1532C00081.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2512&filename=CSR_Synopsis_D1532C00081.pdf